CLINICAL TRIAL: NCT03779646
Title: Bisoprolol for Early Cardiomyopathy in Duchenne Muscular Dystrophy: a Randomized, Controlled Trial
Brief Title: Bisoprolol in DMD Early Cardiomyopathy
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: National Natural Science Foundation of China (Other Government); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Xiaoxiao Guo, Associated professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PekingUMCH-DMD
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Duchenne Muscular Dystrophy; Cardiomyopathy, Dilated
Keywords: Duchenne muscular dystrophy; Early cardiomyopathy; bisoprolol
MeSH Terms: conditions — Muscular Dystrophy, Duchenne; Cardiomyopathy, Dilated; Cardiomyopathies | interventions — Bisoprolol

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled trial.Enrolled participants should receive a kind of ACEI drug for more than 1 month and the dose should be fixed. Then the participants were randomly assigned (1:1) to receive either bisoprolol or not any beta blocker.
Who Masked: Outcomes Assessor
Masking Description: The investigator, care providers and participants will know whether the participants use the trial drug（bisoprolol） or not. But the outcome assessor who will analysis the results of the cardiac MR and echocardiography images from the participants will be blinded to the grouping situation.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bisoprolol fumarate (Experimental): In this arm, the participants will receive different dose of bisoprolol fumarate.
  Interventions: Drug: Bisoprolol Fumarate
- Control (No Intervention): In the control (no beta blocker) group, the patients not taking beta blocker will receive outpatient clinic or video visit every 8 weeks and provide their cardiac symptoms, heart rate, blood pressure and ECG. After 12 months , the patients will repeat cardiac MR besides heart rate, blood pressure, symptoms, ECG,BNP and echocardiography records.

INTERVENTIONS:
Drug: Bisoprolol Fumarate — Bisoprolol was initiated at a dose of 1.25 mg every 24hr. At subsequent biweekly visits, the bisoprolol dose was increased 1.25mg progressively until a daily dose of 0.2mg/kg or the maximum tolerated dose (The rest heart rate <75bpm and systolic blood pressure <90mmHg) is achieved. If the participant feel dizziness or the rest heart rate below 60 bpm or systolic blood pressure below 85mmHg or there is any new onset contraindication to bisoprolol, the doctor will decide to return back to the previous dose or stop bisoprolol. Each time the dose is increased, the medication is administered in an outpatient clinic setting, with assessment of the participant's heart rate, blood pressure, symptoms and ECG. Once reach the target dose, the patients will be followed up every 8 weeks in an face-to-face or video visit. After 12 months , the participants will repeat cardiac MR besides heart rate, blood pressure, symptoms, ECG and brain natriuretic peptide(BNP), echocardiography records.
  Arms: bisoprolol fumarate

SUMMARY:
This study aimed to use cardiac magnetic resonance imaging (CMR) to evaluate the efficacy and safety of bisoprolol therapy for boys with Duchenne muscular dystrophy(DMD) and preserved ejection fraction. On top of angiotensin-converting enzyme inhibitor (ACEI) , half of the participants will receive bisoprolol in combination, while the other half will not receive any beta-blocker.

DETAILED DESCRIPTION:
By the age of 20 years, almost all the patients with Duchenne muscular dystrophy(DMD) have experienced dilated cardiomyopathy (DCM), a condition that contributes significantly to their morbidity and mortality. Studies have shown ACEI to be an effective therapy for DMD boys with early cardiomyopathy. Although bisoprolol has been demonstrated as an effective neurohumoral drug for adult patients with DCM, few data exist concerning its safety and efficacy for the patients with DMD. The investigators hypothesize that the treatment with bisoprolol in addition to background ACEI therapy for 12 months in participants with DMD and early myocardial damage evident with late gadolinium enhancement and preserved ejection fraction, would blunt decline in left ventricular systolic performance.

ELIGIBILITY:
Inclusion Criteria:

* Older than(including) 7 years old
* A definite diagnosis of DMD with muscle pathology confirming the expression of dystrophin lower than 5% and/or confirmed mutations in the DMD gene using a clinical accepted technique that completely defines the mutation.
* Using ACEI or ARB for more than 1 month
* Confirmed myocardial damage in one or more left ventricular segments evident by late gadolinium enhancement and preserved left ventricular systolic function(>45%) by cine cardiac MR in 45 days
* Normal renal function
* Holter and blood pressure shows no contraindication of using bisoprolol

Exclusion Criteria:

* Having metal implanted in body
* Having claustrophobia
* Allergic to gadolinium
* Complicated with other cardiovascular diseases
* Medical history or Holter show bradyarrhythmia like II/III degree atrioventricular block, sick sinus syndrome etc.
* Systolic blood pressure lower than 90mmHg or rest heart rate lower than 75bpm
* Having COPD or asthma history
* Having other complications: tumor, endocrine diseases
* Having beta blockers therapy
* Planned operation in the future 12 months
* Allergic to bisoprolol

Min Age: 7 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2019-01-16 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Calculate the change of left ventricle global longitudinal strain in cardiac MR | baseline and 12 months
  Calculate the change of left ventricle global longitudinal strain in cardiac MR from baseline to 12months for each patients

SECONDARY OUTCOMES:
Calculate the change of left ventricular ejection fraction in cardia MR | baseline and 12 months
  Calculate the change of left ventricular ejection fraction in cardia MR from baseline to 12months for each patients
Calculate the change of ventricle late gadolinium enhancement area in cardia MR | baseline and 12 months
  Calculate the change of ventricle late gadolinium enhancement area in cardia MR from baseline to 12months for each patients
Calculate the change of the level of high-sensitivity cardiac troponin I | baseline and 6months, 12 months
  Calculate the change of the level of high-sensitivity cardiac troponin I from baseline to 6months and 12months for each patients
Calculate the change of the level of NT-proBNP | baseline and 6months, 12 months
  Calculate the change of the level of NT-proBNP from baseline to 6months and 12months for each patients
Calculate the change of E/A ratio assessed by echocardiography | baseline and 12 months
  Calculate the change of diastolic dysfunction (E/A ratio) assessed by echocardiography from baseline to 12months for each patients
Change of the resting heart rate | baseline and 6months, 12 months
  Calculate the change of the resting heart rate from baseline to 6months and 12months for each patients

OTHER OUTCOMES:
Number of participants with All cause mortality, cardiac death, or hospitalized due to heart problem | 12 months
  Number of Subjects with All cause mortality, cardiac death, or hospitalized due to heart problem at the end of study
Number of participants with bisoprolol-related adverse events as assessed by the following definition | 12 months
  Bisoprolol treatment-related adverse events including the dizziness, bradyarrhythmia (resting heart rate lower than 55bpm)，II and III degree atrioventricular block，hypotension

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No